CLINICAL TRIAL: NCT00004852
Title: A Phase II/III 48-Week, Randomized, Double-Blind, Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Lamivudine 300mg Once Daily Vs. Lamivudine 150mg BID in Combination With Zidovudine 300mg BID and Efavirenz 600mg Once Daily in Antiretroviral-Naive Adults With HIV-1 Infection
Brief Title: Safety and Effectiveness of Lamivudine When Given Once a Day Versus Twice a Day in Combination With Other Anti-HIV Drugs in HIV-Infected Adults Who Have Never Received Anti-HIV Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 225D; EPV2000 1
Record Dates: First submitted 2000-03-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-08

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Zidovudine; Drug Administration Schedule; Lamivudine; Genotype; Phenotype; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Efavirenz
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to look at the safety and effectiveness of receiving lamivudine (3TC) once a day versus twice a day as part of an anti-HIV drug combination.

DETAILED DESCRIPTION:
Patients are randomized to receive the same total dosage of 3TC either twice a day (Group 1) or once a day (Group 2) in combination with ZDV and EFV over 48 weeks. Viral load measurements will be performed at Weeks 4, 8, 12, 16, 20, 24, and every 8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 18 years of age or older.
* Are HIV-positive.
* Have a viral load (level of HIV in the blood) of at least 400 copies/ml within 21 days of study entry.
* Have a CD4 count greater than 100 cells/mm3 within 21 days of study entry.
* Agree to practice abstinence or use effective barrier methods of birth control (or, if patient is a woman, unable to have children).

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have taken any antiretroviral (anti-HIV) agent.
* Are pregnant or breast-feeding.
* Are unable to absorb food or have trouble taking medicines by mouth.
* Abuse alcohol or drugs to an extent that may make study participation difficult.
* Are not likely to be able to complete the 48 weeks of study treatment.
* Have a history of pancreatitis (inflamed pancreas) or hepatitis within the last 6 months or any evidence of liver disease.
* Have received an investigational vaccine within the past 3 months or have received gene therapy.
* Have a severe medical condition such as diabetes or heart trouble.
* Have been diagnosed with AIDS.
* Have had radiation therapy or chemotherapy within 30 days of study entry, except for treatment of Kaposi's sarcoma.
* Are taking medications that affect the immune system within 30 days of study entry.
* Are taking medications that may interact with the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09

CONTACTS AND LOCATIONS:
Locations (66):
- United States (46):
  - Phoenix Body Positive, Phoenix, Arizona
  - Pacific Oaks Research, Beverly Hills, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Tower ID Med Associates, Los Angeles, California
  - Davies Med Ctr / c/o HIV Institute, San Francisco, California
  - Kaiser Foundation Hospital, San Francisco, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Bach and Godofsky, Bradenton, Florida
  - TheraFirst Med Ctrs Inc, Fort Lauderdale, Florida
  - North Broward Hosp District, Fort Lauderdale, Florida
  - The Coleman Institute Inc, Fort Lauderdale, Florida
  - The Coleman Institute Inc, Ft. Pierce, Florida
  - Kaiser Permanente Infectious Diseases, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Infectious Disease of Indiana, Indianapolis, Indiana
  - Univ of Kentucky Med Ctr, Lexington, Kentucky
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Boston Med Ctr / Evans - 556, Boston, Massachusetts
  - Antibiotic Research Associates, Kansas City, Missouri
  - East Orange Veterans Administration Med Ctr, East Orange, New Jersey
  - ID Care Inc, New Brunswick, New Jersey
  - ID Care Inc, Princeton, New Jersey
  - ID Care Inc, Randolph Township, New Jersey
  - ID Care Inc, Somerville, New Jersey
  - Albany Med College / Div of HIV Medicine, Albany, New York
  - North Shore Univ Hosp / Div of Infectious Diseases, Manhasset, New York
  - St Vincents Hosp / Clinical Research Program, New York, New York
  - St Lukes / Roosevelt Hosp / HIV Center, New York, New York
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Oklahoma State University / College of Osteopathic Medicine, Tulsa, Oklahoma
  - Associates in Med and Mental Health, Tulsa, Oklahoma
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - Methodist Healthcare, Memphis, Tennessee
  - Univ of Tennessee, Memphis, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Dr David Donnell, Dallas, Texas
  - Nelson-Tebedo Community Clinic, Dallas, Texas
  - Univ of Texas Med Branch, Galveston, Texas
  - Montrose Clinic, Houston, Texas
  - Baylor College of Medicine / Dept of Medicine, Houston, Texas
  - Univ of Texas / Med School at Houston, Houston, Texas
  - Univ of Texas Health Sciences Ctr, San Antonio, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia
- Argentina (2):
  - Hosp Muniz, Buenos Aires
  - CAICI, Rosario - Santa Fe
- Brazil (5):
  - Universidade de Campinas, Campinas - SP
  - Hosp Evandro Chagas Fioernz, Manguinhos RJ
  - Hosp Univ Clementino Fraga Filho, Rio de Janeiro - RJ
  - Hosp Univ Pedro Ernesto / Univ Estadual do RJ, Rio de Janeiro - RJ
  - Hosp Sao Paulo da Universidade Federal de Sao Paulo, Sao Paulo - SP
- Canada (8):
  - Southern Alberta HIV Clinic / Foothills Hosp, Calgary, Alberta
  - Saint Paul's Hosp, Vancouver, British Columbia
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Toronto Gen Hosp, Toronto, Ontario
  - Wellesley/Central Site / St Michael's Hospital, Toronto, Ontario
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
  - Clinique Medicale L'Actuele, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste Foy, Quebec
- Puerto Rico (5):
  - Caguas Regional Hosp, Caguas
  - Hosp San Cristobal-Edif A, Cotto Laurel
  - Carlos Leon-Valiente MD, Guaynabo
  - Ramon Ramirez Ronda MD, Mayagüez
  - San Juan AIDS Program, Santurce